CLINICAL TRIAL: NCT04510142
Title: Questionnaire Follow=up Study Sonia 2
Acronym: QSonia
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Emily Luangrath, Research Nurse, Liverpool University Hospitals NHS Foundation Trust
Other Study IDs: 5870
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Alkaptonuria; Homogentisic Acid; Homogentisate Dioxygenase; Alkaptonuria Severity Score Index
Keywords: Royal Liverpool University Hospital
MeSH Terms: conditions — Alkaptonuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Survey of health of patients completing SONIA 2 study: A cross-sectional analysis by questionnaire

DETAILED DESCRIPTION:
The Liverpool site will post the once only, short questionnaire (in the correct language using translated documents as appropriate) to the address of those patients who completed SONIA 2. Hospital approved translation services will be used. A return-addressed stamped envelope for ease of return will also be provided. Those who received nitisinone will be sent the nitisinone-administration questionnaire and those who did not receive nitisinone will be sent a no-nitisinone questionnaire

ELIGIBILITY:
Inclusion Criteria:

- Documented diagnosis of AKU. Age ≥16 years.

Exclusion Criteria:

- Not completed SONIA 2 study for the full 4-year duration.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cross-sectional cohort who completed SONIA 2 Study
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
to collect information on their health status since completing participation in SONIA 2 | 12 months
  All of the SONIA 2 completed questionnaire data collection is completed by 2 Sept 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Royal Hospitals NHS Foundation Trust, Liverpool, United Kingdom